CLINICAL TRIAL: NCT02944188
Title: Laparoscopic Versus Open Right Hemicolectomy in Treatment of Right-sided Colon Cancer Within an Enhanced Recovery After Surgery (ERAS) Protocol
Brief Title: Laparoscopic Versus Open Right Hemicolectomy Within ERAS in Right-sided Colon Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xu jianmin (Other)
Responsible Party: Sponsor-Investigator, Xu jianmin, Deputy director of the colorectal cancer center, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERAS-02; 82345432 (Other Grant/Funding Number: Shanghai key research projects)
Record Dates: First submitted 2015-07-20; First posted 2016-10-25 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Colon Cancer
Keywords: enhanced recovery after surgery; right hemicolectomy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LRH plus ERAS (Experimental): patients undergo Laparoscopic right hemicolectomy plus ERAS
  Interventions: Procedure: Laparoscopic right hemicolectomy plus ERAS
- ORH plus ERAS (Active Comparator): patients undergo open right hemicolectomy plus ERAS
  Interventions: Procedure: Open right hemicolectomy plus ERAS

INTERVENTIONS:
Procedure: Laparoscopic right hemicolectomy plus ERAS — patients treated with Laparoscopic right hemicolectomy plus enhanced recovery after surgery (ERAS) programs
  Other Names: LRH ERAS
  Arms: LRH plus ERAS
Procedure: Open right hemicolectomy plus ERAS — patients treated Open right hemicolectomy plus enhanced recovery after surgery (ERAS) programs
  Arms: ORH plus ERAS

SUMMARY:
In this study, the investigators have compared the clinical outcomes of the laparoscopic and open right hemicolectomy within enhanced recovery after surgery (ERAS) programs in the treatment of right-sided colon cancer.

DETAILED DESCRIPTION:
This study was a prospective, single-center, randomized control trial. Including criteria were (1) Age between 18 and 75 years; (2) Histologically confirmed right-sided colon adenocarcinoma；(3) Clinical stage I-III; (4) Performance status (ECOG) 0-1; (5) Adequate hematological, hepatic and renal function. Patients operated on as an emergency, or with tumours in the transverse colon, or with other previous malignancy within 5 years were excluded.

All particapants were recruited and randomly assigned to receive laproscopic or open right hemicoloectomy. All patients were treated with an ERAS protocol. The primary end-point was the incidence of postoperative complications within 30 days. Complications were diagnosed and classified according to the Clavien-Dindo classification. The secondary end-points were ERAS adherence, readmissions, reoperations, hospital length of stay, mortality, and survivals. The study was approved by the Ethics Committee of Zhongshan Hospital, Fudan University, Shanghai, China. Written informed consent was obtained for patients to participate the study. This study followed the Consolidated Standards of Reporting Trials (CONSORT) reporting guideline.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years;
2. Primary tumor has undergone histologically confirmed right-sided colon adenocarcinoma;
3. Together with clinical or radiological evidence of Stage(T1-2,N0, M0) Stage II (T3-4, N0, M0) or Stage III (T1-4, N1-2, M0) disease (according to the 2007 revision of the International Union Against Cancer TNM staging system)
4. Performance status (ECOG) 0~1
5. Adequate hematological function: Neutrophils≥1.5 x109/l and platelet count≥100 x109/l; Hb ≥9g/dl (within 1 week prior to randomization)
6. Adequate hepatic and renal function: Serum bilirubin≤1.5 x upper limit of normal (ULN), alkaline phosphatase ≤5x ULN, and serum transaminase (either AST or ALT) ≤ 5 x ULN(within 1 week prior to randomization);
7. Written informed consent for participation in the trial.

Exclusion Criteria:

1. Other previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
2. Pregnancy (absence confirmed by serum/urine β-HCG) or breast-feeding
3. Known drug abuse/ alcohol abuse
4. Legal incapacity or limited legal capacity
5. Pre-existing peripheral neuropathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative complications | 30 days from surgery
  The incidence of postoperative complications within 30 days according to the Clavien-Dindo classification

SECONDARY OUTCOMES:
overall survival | 3 years
  Time from randomization to deaths resulting from any reason
disease-free survival | 3 years
  Time from randomization to recurrence at any site or deaths resulting from any reason
operative mortality | 30 days post operatively
  Deaths related to surgery within 30 days from surgery

OTHER OUTCOMES:
operative time | Day 1
  Time from start of incision to finish of abdomial closure
estimated blood loss | Day 1
  Blood loss will be measured according to the suction and the weight of wet gauze, and then minus the irrigation.
number of retrieved lymph nodes | 1 week post operatively
  Numbers according to the pathological report
postoperative hospital stay | 30 days post operatively
  The postoperative hospital stay is defined as the number of date from the first day after operation to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jiang, MD, Study Director — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China